CLINICAL TRIAL: NCT03776617
Title: Regional Scalp Block With Ropivacaine 0.5% in Patients Undergoing Elective Craniotomy: a Prospective Randomized Controlled Trial
Brief Title: Scalp Block in Elective Craniotomy for Tumor Dissection Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Stachtari Chrysoula MD, PhD, Stachtari Chrysoula, Consultant Anesthesiologist, G. Papanikolaou Hospital, George Papanicolaou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ScalCran
Record Dates: First submitted 2018-05-16; First posted 2018-12-17 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2018-12

CONDITIONS: Craniotomy
Keywords: scalp block; craniotomy; dexmedetomidine; ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group Ropivacaine (Experimental): general anesthesia + scalp block with 20 ml xylocaine 1% and 20ml ropivacaine 0.5%
  Interventions: Procedure: scalp block
- Group Ropivacaine-Dexmedetomidine (Experimental): general anesthesia + scalp block with 20 ml xylocaine 1%, 20ml ropivacaine 0.5% and 1mcg/kg dexmedetomidine
  Interventions: Procedure: scalp block
- Group control (No Intervention): general anesthesia
- Group sham (Sham Comparator): general anesthesia + Scalp block with 40ml Normal Saline
  Interventions: Procedure: scalp block

INTERVENTIONS:
Procedure: scalp block — Scalp block will be performed five minutes before head pinning for elective craniotomy by blocking supraorbital, auriculotemporal, occipital and postauricular branches of the greater auricular nerves.
  Arms: Group Ropivacaine; Group Ropivacaine-Dexmedetomidine; Group sham

SUMMARY:
This study was designed to evaluate the effect of scalp block combined with general anesthesia on the intraoperative consumption of fentanyl and time of extubation of patients undergoing elective craniotomy. Scalp block will be applied to three groups with differences of the administered solution to the scalp and one group will be placebo group.

DETAILED DESCRIPTION:
Regional scalp block (RSB) is an established technique that involves infiltration of local anesthetic (LA) at well-defined anatomical sites targeting the major sensory innervation of the scalp. Regional techniques minimize anesthetic requirements and their effects may be beneficial. There is a lack of consensus and evidence concerning alternative analgesia strategies for cranial neurosurgery.

Patients undergoing elective craniotomy for tumor dissection will be randomly divided into four groups to receive scalp block as an adjuvant to general anesthesia. After a standard induction sequence using propofol, fentanyl and a single dose of rocuronium, patients will be intubated. Bilateral scalp block will be given immediately after induction, except patients in control group who will not have a scalp block. Drugs for scalp block will be 20ml ropivacaine 0.5%, 20ml xylocaine 1% and dexmedetomidine 1mcg/kg.Anaesthesia will be maintained with propofol and remifentanyl infusion. Intraoperatively, propofol infusion at 75 to 100 μg/kg/h up to dura closure and reduced to 50-75 μg/kg/h up to skin closure. Five minutes before head pinning scalp block was performed by blocking the supraorbital, supratrochlear, auriculotemporal, occipital, and postauricular branches of the greater auricular nerves.Routine monitoring of electrocardiogram, heart rate (HR), and mean arterial blood pressure (MAP) will record at two-minute intervals from the beginning of anesthesia until 10 minutes after incision, followed by 5-minute intervals throughout the remaining course of the surgery. Monitoring of the depth of anesthesia will also performed using the Bispectral Index. Sample size was calculated based on Type I error of α = 5% and power = 80% and minimum difference d = 30%, which is clinically significant in the pilot study. All quantitative variables will be reported as mean and standard deviation, and qualitative variables will be listed as number (percentage). Mann-Whitney test and Chi-square test will be used for comparison of endpoints. Linear mixed model will be used to evaluate the differences of hemodynamics variables. Statistical Package for Social Sciences (SPSS, version 19.0; SPSS Inc., Chicago, USA) will be used for all calculations. p values less than .05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists Physical status classification 1-3
* patients who are scheduled for elective craniotomy for brain tumor
* patients who have provided consent for participation in the study

Exclusion Criteria:

* Patients who have allergy to local anesthetics and dexmedetomidine
* Glasgow coma scale <15
* tumor>4cm
* any contraindication for receiving dexmedetomidine
* severe mental impairment
* pregnant women
* uncontrolled hypertension, arrhythmia, coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
intraoperative opioid consumption | intraoperative
  The overall intravenous fentanyl and remifentanil consumption (microgram/ kilogram) during the surgery. The decision to administer fentanyl is guided by the changes of blood pressure and/ or heart rate greater than 20% from baseline level.
systolic arterial pressure and diastolic arterial pressure | intraoperative
  The systolic and diastolic blood pressure and heart rate change from baseline will be calculated. The unit for blood pressure is mmHg.
heart rate fluctuation | intraoperative
  heart rate change from baseline will be calculated. The unit for heart rate is bpm

SECONDARY OUTCOMES:
extubation time | one day
  Time from the end of anesthetic to fully awake and extubation

OTHER OUTCOMES:
chronic pain after craniotomy | 3 months after craniotomy
  telephone after 3 months and ask for pain description using the Numeric Pain Rating Scale (NPRS). A respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Trikoupi, MD, PhD, Study Director — General Hospital of Thessaloniki
Locations (1):
- George Papanikoalou Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No